CLINICAL TRIAL: NCT05058001
Title: Accuracy of Prenatal Ultrasonography in The Diagnosis Of Neurological Fetal Anomalies
Brief Title: Diagnosis Of Neurological Fetal Anomalies
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Bothina Zakria Elsayed, Assistant lecturer, Sohag University
Other Study IDs: Soh-Med-21-09-21
Record Dates: First submitted 2021-09-10; First posted 2021-09-27 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Fetal Anomaly of Central Nervous System
Keywords: Sonography ,neurlogical anomalies

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a descriptive cross-sectional study 300 patients coming for antenatal care at sohag governorate undergo mid anatomical scan.

Samples 300 pregnant women have mid anatomical scan at 20-22 weeks as routine antenatal care and Examination of the fetal CNS will be performed with a high resolution two dimensional ultrasound machine (Voluson E8) equipped with a RAB 4 to 8MHz multifrequency transabdominal Probe. Four standard recommended views-transventricular, falx, cavum, and posterior fossa or transcerebellar views-provide an overview of fetal intracranial anatomy during the second trimester anatomy scan.

Follow-up information will be obtained in all cases, and all infants will be considered healthy by pediatric examination. In selected cases, postnatal single-shot fast spin-echo magnetic resonance (MR) imaging will be performed as integrated, complementary investigation.to confirm diagnosis.

DETAILED DESCRIPTION:
1. Type of the study: This is a descriptive cross-sectional study
2. Study Setting: 300 patients coming for antenatal care at sohag governorate undergo routine second trimester scan.
3. patients and methods:

Inclusion criteria:

1. All pregnant females of 18 to 45 years old.
2. gestational age of 20- 22 gestational week .

Exclusion criteria:

1-age less than18years and more than 45 years. gestational age less or more than20- 22 weeks. Samples Methods 300 pregnant women low risk pregnancy will be scanned at 20-22 weeks as routine antenatal care and Examination of the fetal CNS will be performed with a high resolution two dimintional ultrasound machine (Voluson E8) equipped with a RAB 4 to 8MHz multifrequency transabdominal Probe. Four standard recommended views-transventricular, falx, cavum, and posterior fossa or transcerebellar views-provide an overview of fetal intracranial anatomy during the second trimester anatomy scan.

Follow-up information will be obtained in all cases, and all infants will be considered healthy by pediatric examination. In selected cases, postnatal single-shot fast spin-echo magnetic resonance (MR) imaging will be performed as integrated, complementary investigation.to confirm diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant females of 18 to 45 years old.
* gestatioal age of 20- 22 gestational week .

Exclusion Criteria:

* age less than18years and more than 45 years.
* gestational age less or more than20- 22 weeks.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Study Population: 300 pregnant women have mid anatomical scan at 20-22 weeks as routine antenatal care and Examination of the fetal CNS will be performed with a high resolution two dimintional ultrasound machine (Voluson E8) equipped with a RAB 4 to 8MHz multifrequency transabdominal Probe.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Accuracy of sonography in the diagnosis of neurological fetal anomalies | From 20 _ 22 gestational age ...confirmation occursat birth till 1 week post natal
  Investigator compares the accuracy of songraphy in the diagnosis of neurological fetal anomalies with post natal diagnosis by either clinically or by MRIThis is a descriptive cross-sectional study 2- Study Setting: 300 patients coming for antenatal care at sohag governorate undergo mid anatomical scanExamination of the fetal CNS will be performed with a high resolution two dimintional ultrasound machine (Voluson E8) equipped with a RAB 4 to 8MHz multifrequency transabdominal Probe. Four standard recommended views-transventricular, falx, cavum, and posterior fossa or transcerebellar views-provide an overview of fetal intracranial anatomy during the second trimester anatomy scan.
  After birth ,investigator reports anomalies clinically or after consultation of pediatric department.

CONTACTS AND LOCATIONS:
Overall Officials: Bothyna Za Elsayed, Assistant lecturer, Principal Investigator — Sohag University
Locations (1):
- Medicine, Sohag, Sohag Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No